CLINICAL TRIAL: NCT02305264
Title: Imaging of Intracerebral Inflammation in the Progressive Phase of Multiple Sclerosis
Brief Title: Imaging of Intracerebral Inflammation in MS
Acronym: INFLASEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P091001
Record Dates: First submitted 2013-01-25; First posted 2014-12-02 (Estimated); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive; Multiple Sclerosis, Primary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET -18F-DPA-714 and 18F-FDG (Experimental): 18F-DPA-714, dose 5mCi (185MBq), will be injected via an arm intravenous catheter.
  18F-FDG , dose 5mCi(185MBq), will be injected via an arm intravenous catheter.
  Interventions: Drug: 18F-DPA-714 and 18F-FDG

INTERVENTIONS:
Drug: 18F-DPA-714 and 18F-FDG — Positron emission tomography (PET) imaging following the injection of 2 radiotracers (here considered as the drugs): 1) 18F-DPA-714 ii) 18F-FDG. PET -18F-DPA-714, dose 5mCi (185MBq), will be injected via an arm intravenous catheter.
  18F-FDG , dose 5mci(185MBq), will be injected via an arm intravenous catheter.

SUMMARY:
In this study we plan to image the compartmentalized inflammation in MS using molecular imaging by positron emission tomography (PET) with a very highly resolutive camera. Two tracers will be studied and compared: i) [18F]DPA-714, which bind to the peripheral benzodiazepine receptor (PBR), a target mainly expressed by activated microglial cells. This new ligand for PBR displays several advantages compared to the existing reference compound PK11195 in term of brain entrance, signal to noise ratio, and radiolabelling possibility with [18F] ii) [18F]-fluoro-desoxy-glucose ([18F]FDG), which should reflect glucose metabolism in activated immune cells in the white matter. Progressive MS patients (secondary progressive and primary progressive) will be compared to relapsing-remitting patients and to healthy volunteers. All subjects will pass a complete neurological evaluation and a multimodal MRI to document clinical disability and tissue injury. A clinical and radiological follow up will then be performed for a 2-year period. This study should help to understand the contribution of the intracerebral inflammation on the progression of disability and could provide a surrogate marker for further therapeutic trials in chronic progressive MS.

DETAILED DESCRIPTION:
Study design This study is a prospective cross-sectional controlled multicentric clinical study in 45 MS patients and 20 controls.

Four groups of person will be included and compared:

* Group I: 20 healthy volunteers aging from 18 to 65 years. These healthy volunteers will be matched for age and sex with patients (1/2).
* Group II: 15 patients aging from 18 to 65 years with relapsing-remitting (RRMS), with less than 10 years of evolution since the first manifestation and no recent relapse.
* Group III: 15 patients aging from 18 to 65 years with secondary progressive MS (SPMS), with less than 10 years of evolution since the occurrence of the secondary progressive phase.
* Group III: 15 patients aging from 18 to 65 years with primary progressive MS (PPMS) diagnosed since less than 10 years.

Study centres MS patients and the 20 healthy volunteers will be recruited in the Hospital Pitie-Salpetriere

MS patients will be recruited in the Hospital Tenon

This study will be performed by complementary teams already collaborating on molecular imaging trials in MS (which assess neuronal loss or demyelination/remyelination): i) the "Centre d'Investigation Clinique" (Salpetriere hospital, Paris), which is strongly experienced in the coordination of clinical and translational research on MS; ii) the CENIR (centre for neuroimaging research, Salpetriere hospital, Paris) a specialized MRI centre for research on neurological diseases; iii) the SHFJ (DSV, CEA, ORSAY) which is a world class molecular imaging centre;

Study duration Per patient the study will last two years Per control the study will last up to 8 weeks

ELIGIBILITY:
Inclusion criteria

Healthy volunteers (group I, n=20)

* Aged 18-65 years;
* Able to understand the objectives and procedures of the study, and who give inform consent.

Patients with relapsing-remitting MS (group II, n=15)

* Aged 18-65 years
* Clinically definite MS according to McDonald revised criteria
* Less than 10 year of evolution
* No clinical relapse during the past 3 months
* Able to understand the objectives and procedures of the study, and who give inform consent

Patients with progressive MS (group III and IV, n=15 per group)

* Aged 18-65 years
* Clinically definite MS according to McDonald revised criteria
* SPMS evolving since more than 10 years for group III (n = 15).
* PPMS evolving since less than 10 years for group IV (n=15).
* Each progressive patient should have experienced a significant progression during the 2 years preceding the inclusion (with an estimated progression of the EDSS score of at least 0.5 point).
* No clinical relapse during the past 3 months
* Able to understand the objectives and procedures of the study, and who give inform consent.

Exclusion criteria

* Any reason, which does not allow performing MRI: claustrophobia, pace-maker or intra-ocular foreign body for example.
* For women: pregnancy, lactation, lack of efficient contraception. At visit 2, a positive pregnancy test will lead to exclude the patient.
* Uncontrolled diabetes
* Current symptoms of severe or uncontrolled renal, hepatic, hematological, gastrointestinal pulmonary or cardiac disease.
* Positive HIV test
* Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual guidelines.
* Other chronic neurological disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-03-19 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Whole brain Binding Potential (BP) of 18F-DPA-714 | D0
  Quantification of microglial compartmentalized inflammation within the brain by PET with 18F-DPA-714 in MS patients and healthy controls

SECONDARY OUTCOMES:
Binding potential of 18F-DPA-714 in segmented brain regions | D0
  To compare binding potential of 18F-DPA-714 in segmented brain regions: white matter, gray matter, white matter lesions
Binding potential of 18F-DPA-714 in subgroups of MS patients | D0
  To compare binding potential of 18F-DPA-714 in subgroups of MS patients (secondary progressive, primary progressive, relapsing remitting)
Predictive value of PET 18F-DPA-714 BP on neurological clinical metrics | 2 years
  To determine the predictive value of brain microglial inflammation on subsequent neurological impairment progression after a follow up period of two years.
Predictive value of PET 18F-DPA-714 BP on MRI metrics | 2 years
  To determine the predictive value of brain microglial inflammation on subsequent brain atrophy progression after a follow up period of two years.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Stankoff, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Saint Antoine Hospital, Paris
  - Pitie Salpetriere Hospital, Paris

REFERENCES:
- [Derived] Peyronneau MA, Kuhnast B, Nguyen DL, Jego B, Sayet G, Caille F, Lavisse S, Gervais P, Stankoff B, Sarazin M, Remy P, Bouilleret V, Leroy C, Bottlaender M. [18F]DPA-714: Effect of co-medications, age, sex, BMI and TSPO polymorphism on the human plasma input function. Eur J Nucl Med Mol Imaging. 2023 Sep;50(11):3251-3264. doi: 10.1007/s00259-023-06286-1. Epub 2023 Jun 9. PMID 37291448
- [Derived] Ricigliano VAG, Louapre C, Poirion E, Colombi A, Yazdan Panah A, Lazzarotto A, Morena E, Martin E, Bottlaender M, Bodini B, Seilhean D, Stankoff B. Imaging Characteristics of Choroid Plexuses in Presymptomatic Multiple Sclerosis: A Retrospective Study. Neurol Neuroimmunol Neuroinflamm. 2022 Oct 13;9(6):e200026. doi: 10.1212/NXI.0000000000200026. Print 2022 Nov. PMID 36229188
- [Derived] Garcia-Lorenzo D, Lavisse S, Leroy C, Wimberley C, Bodini B, Remy P, Veronese M, Turkheimer F, Stankoff B, Bottlaender M. Validation of an automatic reference region extraction for the quantification of [18F]DPA-714 in dynamic brain PET studies. J Cereb Blood Flow Metab. 2018 Feb;38(2):333-346. doi: 10.1177/0271678X17692599. Epub 2017 Feb 9. PMID 28178885